CLINICAL TRIAL: NCT05637294
Title: Effect of Night-time and Full-time Splinting for Carpal Tunnel Syndrome: a Multi-center, Three-period, Randomized Cross-over Superiority Trial (FINCROSS - Finnish Crossover Trial for Carpal Tunnel Syndrome)
Brief Title: Effect of Night-time and Full-time Splinting for Carpal Tunnel Syndrome
Acronym: FINCROSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Terveystalo (Other); Hospital Nova of Central Finland (Unknown); Mikkeli Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R22093
Record Dates: First submitted 2022-10-18; First posted 2022-12-05 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; splinting; no-treatment; cross-over trial
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Splints

STUDY DESIGN:
Intervention Model Description: Multicentre, three-treatment, three-period, randomised, crossover superiority trial (3 x 6 crossover design)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence of three treatment periods in the following order: ABC (Other): Splinting at night while sleeping for 6 weeks (period A), then no treatment for 6 weeks (period B), then splinting at day and night for 6 weeks (period C). Each treatment period will be separated by 3-week washout period.
  Interventions: Device: splinting
- Sequence of three treatment periods in the following order: ACB (Other): Splinting at night while sleeping for 6 weeks (period A), then splinting at day and night for 6 weeks (period C), then no treatment for 6 weeks (period B). Each treatment period will be separated by 3-week washout period.
  Interventions: Device: splinting
- Sequence of three treatment periods in the following order: BAC (Other): No treatment for 6 weeks (period B), then splinting at night while sleeping for 6 weeks (period A), then splinting at day and night for 6 weeks (period C). Each treatment period will be separated by 3-week washout period.
  Interventions: Device: splinting
- Sequence of three treatment periods in the following order: BCA (Other): No treatment for 6 weeks (period B), then splinting at day and night for 6 weeks (period C), then splinting at night while sleeping for 6 weeks (period A). Each treatment period will be separated by 3-week washout period.
  Interventions: Device: splinting
- Sequence of three treatment periods in the following order: CAB (Other): Splinting at day and night for 6 weeks (period C), then splinting at night while sleeping for 6 weeks (period A), then no treatment for 6 weeks (period B). Each treatment period will be separated by 3-week washout period.
  Interventions: Device: splinting
- Sequence of three interventions/treatments in the following order: CBA (Other): Splinting at day and night for 6 weeks (period C), then no treatment for 6 weeks (period B), then splinting at night while sleeping for 6 weeks (period A). Each treatment period will be separated by 3-week washout period.
  Interventions: Device: splinting

INTERVENTIONS:
Device: splinting — neutral-positioned wrist orthosis

SUMMARY:
Carpal tunnel syndrome is a common compression neuropathy of upper extremities. Its usual symptoms are pain, numbness and tingling of fingers, which tend to be worse at night. Splinting the wrist with an external orthosis is usually a first-line treatment provided to most people with mild to moderate disease.

The FINCROSS trial (randomized cross-over trial) aims to assess the effect of night-time and full-time splinting in comparison with no-treatment. It also aims to identify possible subgroups of people who would benefit from splinting, as well as assess if positive response to splinting is associated with subsequent lower need of surgery.

The trial will recruit 110 people with carpal tunnel syndrome in Finland. Each participant will undergo all three treatment periods in a randomised order: 1) splinting at night-time for six weeks, 2) splinting both day and night for six weeks; and 3) be assessed under a six weeks long control period of no-treatment.

Each treatment period will be separated with a three-week washout period. Therefore, the whole treatment sequence for each participant lasts 24 weeks after randomization. The participant will be followed-up to 1 year after the randomisation.

Additionally, the participants will get instructions for self-administered stretching exercises to perform throughout the study. All participants will be asked to avoid any intervention administered or supervised by medical personnel (such as structured supervised exercises, manual therapy, steroid injections, surgery, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Clinically confirmed carpal tunnel syndrome (CTS) of any severity level (diagnostic criteria: numbness, pain or paraesthesia in the median nerve distribution area of wrist and fingers),
2. Symptom duration of CTS for at least 3 weeks,
3. No previous corticosteroid injection for CTS during last 6 months,
4. No previous surgery for CTS,
5. Aged 18 years or older,
6. Able to complete self-report questionnaires electronically,
7. Able to understand Finnish,
8. Willing to join the study and follow the study protocol instructions,
9. Sign informed consent.

Exclusion Criteria:

1. Nerve root or plexus disorders that might be causing CTS mimicking symptoms (e.g., cervical radiculopathy, thoracic outlet syndrome, or whiplash associated disorders),
2. Other neurological condition affecting the function of the hand such as Multiple Sclerosis, previous nerve injury,
3. Active Rheumatoid arthritis or any other active inflammatory joint disease affecting the hand,
4. Thenar muscle atrophy,
5. Untreated hypothyroidism,
6. Known allergy to any of the splint materials (self-reported by patient),
7. Long term treatment (over 4 months) for CTS with no response,
8. Any other known reason that could prevent from participation for the study time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change of The 6-item CTS Symptoms Scale scores between baseline and 6 weeks | 6 weeks, i.e. end of each treatment period
  6-item CTS Symptoms Scale is a 6-item questionnaire, with score from 1 to 5 to each of the item, higher score indicating worse symptoms. The study will use a Finnish version of The 6-item CTS Symptoms Scale.

SECONDARY OUTCOMES:
Change of The 6-item CTS Symptoms Scale scores between baseline and 3 weeks | 3 weeks, i.e. middle of each treatment period
  6-item CTS Symptoms Scale is a 6-item questionnaire, with score from 1 to 5 to each of the item, higher score indicating worse symptoms. The study will use a Finnish version of The 6-item CTS Symptoms Scale.
Change of The 6-item CTS Symptoms Scale scores between baseline and 1 year | 1 year
  6-item CTS Symptoms Scale is a 6-item questionnaire, with score from 1 to 5 to each of the item, higher score indicating worse symptoms. The study will use a Finnish version of The 6-item CTS Symptoms Scale.
Change of The Boston Carpal Tunnel Questionnaire Symptom Severity Scale scores (BCTQ SSS) between baseline and 6 weeks of each treatment period | 6 weeks, i.e. end of each treatment period
  BCTQ SSS is an 11-item questionnaire, with score from 1 to 5 to each of the item, higher score indicating worse symptoms. The study will use a Finnish version of the BCTQ SSS.
Change of The Boston Carpal Tunnel Questionnaire Symptom Severity Scale scores (BCTQ SSS) between baseline and 1 year | 1 year
  BCTQ SSS is an 11-item questionnaire, with score from 1 to 5 to each of the item, higher score indicating worse symptoms. The study will use a Finnish version of the BCTQ SSS.
Change of The Boston Carpal Tunnel Questionnaire Functional Status Scale (BCTQ FSS) between baseline and 6 weeks of each treatment period | 6 weeks, i.e. end of each treatment period
  BCTQ FSS is an 8-item questionnaire, with score from 1 to 5 to each of the item, higher score indicating worse function. The study will use a Finnish version of the BCTQ FSS.
Change of The Boston Carpal Tunnel Questionnaire Functional Status Scale (BCTQ FSS) between baseline and 1 year | 1 year
  BCTQ FSS is an 8-item questionnaire, with score from 1 to 5 to each of the item, higher score indicating worse function. The study will use a Finnish version of the BCTQ FSS.
Change of The Boston Carpal Tunnel Questionnaire (BCTQ) Total between baseline and 6 weeks | 6 weeks, i.e. end of each treatment period
  BCTQ Total consists of BCTQ SSS and BCTQ FSS, with score from 1 to 5 to each of the item, higher score indicating worse function.
Change of The Boston Carpal Tunnel Questionnaire (BCTQ) Total between baseline and 1 year | 1 year
  BCTQ Total consists of BCTQ SSS and BCTQ FSS, with score from 1 to 5 to each of the item, higher score indicating worse function.
Overall improvement as measured by 7-point Likert Scale | 6 weeks, i.e. end of each treatment period
  7-point Likert Scale assesses the improvement of hand symptoms with 7 possible scores: much better, better, somewhat better, no changes, somewhat worse, worse, much worse.
Overall improvement as measured by 7-point Likert Scale | 1 year
  7-point Likert Scale assesses the improvement of hand symptoms with 7 possible scores: much better, better, somewhat better, no changes, somewhat worse, worse, much worse.
Change of The EuroQol 5-dimension (EQ-5D-5L) Health Status and Quality-of-life Measure score between baseline and 6 weeks of each treatment period | 6 weeks, i.e. end of each treatment period
  Finnish version of EQ-5D-5L will be used.
Change of The EuroQol 5-dimension (EQ-5D-5L) Health Status and Quality-of-life Measure score between baseline and 1 year | 1 year
  Finnish version of EQ-5D-5L will be used.
Adverse effects | up to 1 year
  Assessed by participant self-reported adverse events.
Need for surgery | up to 1 year
  Assessed by participant self-reported information of referral to or executed surgery.
Escape treatments (e.g., corticosteroid injection or any other treatment supervised by medical personnel) | up to 1 year
  Assessed by participant self-reported information of undergoing or having undergone the escape treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Teemu Karjalainen, Principal Investigator — Tampere University Hospital; Jarkko Jokihaara, Principal Investigator — Tampere University Hospital
Locations (6):
- Finland (6):
  - Terveystalo Kamppi, Helsinki
  - Hospital Nova of Central Finland, Jyväskylä
  - Terveystalo Jyväskylä, Jyväskylä
  - Mikkeli Central Hospital, Mikkeli
  - Tampere University Hospital, Tampere
  - Terveystalo Tampere, Tampere

IPD SHARING:
Plan to Share IPD: No